CLINICAL TRIAL: NCT01437293
Title: Behavioral and Physiological Effects of Cocaine in Cocaine-dependent Participants Treated With Levodopa in Combination With Carbidopa and Entacapone (LCE)
Acronym: COST
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, National Institute on Drug Abuse (NIDA)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: #6141 P50 DA 009236-16; P50DA009236 (NIH); P50DA009236-16 (NIH)
Record Dates: First submitted 2010-11-18; First posted 2011-09-20 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Abuse
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Levodopa; Carbidopa; entacapone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): L-dopa / carbidopa / entacapone (LCE)
  Interventions: Drug: L-dopa / carbidopa / entacapone (LCE)

INTERVENTIONS:
Drug: L-dopa / carbidopa / entacapone (LCE) — For this trial we propose a target dosage of L-dopa / carbidopa / entacapone of 400 mg L-dopa / 100mg carbidopa / 200 mg entacapone, twice daily.
  Other Names: L/C/E

SUMMARY:
An inpatient safety study to characterize the cardiovascular and behavioral effects of cocaine administration in the presence of LCE. The proposed study involves an inpatient stay of 12 days during which participants will have two cocaine-administration sessions, each including five doses of smoked cocaine with ascending doses.

DETAILED DESCRIPTION:
Cocaine dependence remains a serious public health problem; however no clearly effective pharmacological treatments have been identified to date. We hypothesize that identification of subgroups of cocaine-dependent patients will help to develop targeted and more effective treatments. We hypothesize that individuals who have difficulties in achieving abstinence have a deficit in dopaminergic functioning and correcting this deficit using dopaminergic medication levodopa in combination with carbidopa and entacapone (LCE) to increase availability and uptake of levodopa to synthesize dopamine in the brain will result in clinical improvement. We were unable to locate any clinical reports that might provide data on the interaction between cocaine and LCE. Therefore, we would like to conduct an inpatient safety study to characterize the cardiovascular and behavioral effects of cocaine administration in the presence of LCE. The proposed study involves an inpatient stay of 12 days during which participants will have two cocaine-administration sessions, each including five doses of smoked cocaine with ascending doses. Participants will be maintained on placebo capsules prior to the first study session and on the LCE prior to the second session. Physiological (HR, BP, ECG) as well as behavioral (subjective effects) effects of cocaine will be monitored during cocaine-administration sessions. Serial blood samples will also follow cocaine administration to assess whether the pharmacokinetics of cocaine is altered during treatment with LCE. All participants will also undergo two cognitive testing sessions, one on placebo and one on LCE, employing a computerized battery (Quarters, Gambling task, Drug Stroop, Threat Responsivity task). There will be an optional functional MRI (fMRI) component that will investigate behavioral and neural indicators of reward responsivity, thought to reflect dopaminergic transmission. Participants choosing to undergo fMRI testing will complete two sessions, on the same days as the cognitive task sessions. Data obtained in the present study will be used to inform the large, controlled trial of LCE in treatment seeking cocaine-dependent individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 21-50.
* Smokes cocaine on average at least 1x/week; currently spends at least $30/week on cocaine. Has been using cocaine for at least 6 months Urine toxicology positive for cocaine metabolites
* Has patterns of smoked cocaine use in terms of frequency and amount that parallels or exceed those administered in the study
* Able to give informed consent and comply with study procedures

Exclusion Criteria:

* Current DSM-IV criteria of substance use disorders with the exception of cocaine or nicotine dependence, or a history of alcohol or cannabis dependence.
* Request for drug treatment
* Unstable medical disorders, or medical disorders that might interfere with study participation, including current seizure disorder, heart disease or a history of serious adverse effects due to cocaine.
* Judged to be noncompliant with study protocol
* Concurrent use of any psychotropic medications
* Concurrent use of MAO inhibitors or epinephrine (patients must be off MAOIs for a minimum of 2 weeks)
* Clinical laboratory tests outside normal limits that are clinically unacceptable to the study physician (systolic BP > 140 and < 90, diastolic BP > 90 and < 60, and heart rate > 90; BUN, creatinine, LFTs > ULN; hematocrit < 34 for women, < 36 for men; pseudocholinesterase deficiency)
* Positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control
* History of myocardial infarction or ischemia, clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse
* History of narrow angle glaucoma or prostate cancer
* History of melanoma or current suspicious undiagnosed skin lesions
* Currently meeting DSM-IV criteria for all major psychiatric/psychotic disorders other than transient psychosis due to drug abuse
* History of allergic reaction or adverse reaction to study medications (levodopa/carbidopa/entacapone).
* Current parole or probation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure | (baseline) prior to and after each of the 6 cocaine administrations at 4, 18, 32, 46, 60, 74, 104 and 134 minutes after the first dose
  Maximum SBP, maximum DPB will be obtained at baseline, prior to the first session dose, and after each consecutive dose (0, 6, 12, 25, 50, 50 mg). Changes from baseline in blood pressure in the used by cocaine administration under placebo condition will be compared to those obtained during treatment with LCE using repeated measures ANOVA.
heart rate | (baseline) prior to and after each of the 6 cocaine administrations at 4, 18, 32, 46, 60, 74, 104 and 134 minutes after the first dose
  Heart rate will be obtained at baseline, prior to the first session dose, and after each consecutive dose (0, 6, 12, 25, 50, 50mg). Changes from baseline in heart rate in the used by cocaine administration under placebo condition will be compared to those obtained during treatment with LCE using repeated measures ANOVA.

SECONDARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | 18, 32, 46, 60, 74, 104 minutes post dose
  Cmax, Area Under Curve, Tmax
subjective cocaine experience | Done at baseline and at 4, 18, 32, 46, 60, 74, 104 and 134 minutes after the first dose
  1) An assessment of the subjective cocaine experience with and without study medication using a standard battery of 100 mm visual analog scales (VAS) that will be administered pre-dosing and after each dose. Each VAS item will be summarized using AUC, mean and peak scores collected for all time points and analyzed using ANOVA with corrections for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: stars website — http://stars.columbia.edu